CLINICAL TRIAL: NCT07025291
Title: Evaluation of Salivary Hypoxia-Inducible Factor -2 Alpha, Matrix Metalloproteinase-9 and Tartrate-Resistant Acid Phosphatase-5b Levels in Individuals With Different Periodontal Diseases
Brief Title: Assessment of Salivary Biomarker Levels in Individuals With Various Periodontal Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Beril Aktan, Research Assistant, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-SAEK-0421
Record Dates: First submitted 2025-06-10; First posted 2025-06-17 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Periodontal Diseases
Keywords: periodontitis; gingivitis; saliva; HIF-2a; TRAP-5b; MMP-9; ELISA
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Gingivitis; Erythrocytosis, Familial, 4

STUDY DESIGN:
Intervention Model Description: According to full-mouth clinical periodontal measurements including probing depth (PD), clinical attachment level (CAL),bleeding on probing (BOP), gingival index (GI) and plaque index (PI) samples of saliva were obtained from 60 systemically healthy non-smoker individuals with periodontitis (P, n=20), gingivitis(G, n=20) and healthy periodontium (S, n=20).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- healthy periodontium (Experimental): According to the evaluation made in 6 areas of each tooth, 20 individuals who showed bleeding on probing in less than 10% of the area, had a probing depth of less than 4 mm and had no attachment loss will be included in the study.
  Interventions: Diagnostic Test: saliva obtaining
- Gingivitis (Experimental): According to the evaluation made in 6 areas of each tooth, 20 individuals who showed bleeding on probing in more than 10% of the area, had a probing depth of less than 4 mm and had no attachment loss will be included in the study.
  Interventions: Diagnostic Test: saliva obtaining
- periodontitis (Experimental): According to the evaluation made in 6 areas of each tooth, 20 individuals who showed bleeding on probing in 30% or more areas, who had a probing pocket depth of 5 mm or more and attachment loss of 4 mm or more in at least 2 non-adjacent teeth in each quadrant jaw, and who had coronal 1/3 or more (horizontal and/or vertical) bone loss on radiographs will be included in the study.
  Interventions: Diagnostic Test: saliva obtaining

INTERVENTIONS:
Diagnostic Test: saliva obtaining — The patient was asked to sit upright and tilt his/her head forward to collect saliva samples. İn this way, unstimulated saliva was allowed to accumulate in the floor of the mouth. The accumulated salivav was collected in a sterile container. It was then transferred to a propylene tube. The tubes were centrifuged and the clear part at the top of the tube was taken with a sterile syringe and transferred to a different propylene tube with 0.5 ml in each tube. Tubes were stored at -80ºC until the day of analysis.

SUMMARY:
The aim of this study is to compare the salivary levels of HIF-2 alpha, MMP-9, and TRAP-5b among healthy individuals, patients with gingivitis, and patients with periodontitis; to examine the relationship between these levels and clinical parameters; and to determine their effectiveness in distinguishing periodontal disease from a healthy condition. It will be evaluated whether these biochemical mediators can be used as diagnostic biomarkers in the diagnosis of periodontal disease.

Periodontal health is defined as the absence of signs of inflammation. Gingivitis is an inflammation of the gums and, if left untreated, can progress to periodontitis, a more severe condition characterized by the destruction of the supporting structures of the teeth. In this destruction, the host immune response to bacterial products and various inflammatory mediators (cytokines, MMPs) play a role.

MMP-9 plays a significant role in the progression of inflammation and tissue damage. HIF-2 alpha is a factor that regulates bone formation and resorption and is activated in hypoxic or inflammatory environments. TRAP-5b is a specific marker of osteoclast activity and bone resorption. In the literature, there is no study that evaluates these three biomarkers together in saliva samples in the context of periodontal disease.

This study aims to investigate the changes in these salivary biomarkers in the presence of periodontal disease, their diagnostic potential, and their relationship with clinical parameters. The findings may also provide insights for future treatments targeting these cytokine pathways.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy (The identification of healthy volunteers will be based on patients' self-reported medical history; no additional diagnostic tests will be conducted.)
* Having at least twenty permanent teeth in the mouth
* Non-smoker
* Not on any continuous medication
* No use of antibiotics, anti-inflammatory drugs, or systemic corticosteroids in the last 6 months
* Not pregnant or lactating
* No periodontal treatment within the last 6 months
* Willing to participate in the study and having signed the "Informed Consent Form"
* Between 18 and 70 years of age

Exclusion Criteria:

* Having any oral or systemic disease
* Being on regular systemic medication
* Being pregnant or in the lactation period
* Having received periodontal treatment within the last 6 months
* Having used antibiotics, anti-inflammatory drugs, or systemic corticosteroids in the last 6 months
* Smoking
* Being under 18 years of age

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-10-10 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Salivary HIF-2α levels | 24 hours after taking the clinical measurements at the first visit
  the total amount of HIF-2α in saliva
Salivary TRAP-5b levels | 24 hours after taking the clinical measurements at the first visit
  the total amount of TRAP-5b in saliva
Salivary MMP-9 levels | 24 hours after taking the clinical measurements at the first visit
  the total amount of MMP-9 in saliva

SECONDARY OUTCOMES:
probing depth | During the first 1 day visit
  With the help of a periodontal probe, the distance between the gingival margin and the sulcus/pocket base will be measured from six points of the tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatinal/lingual, mid buccal/palatinal and distobuccal/palatinal. During the measurement, care will be taken to ensure that the probe is parallel to the long axis of the tooth and that excessive force is not applied. The values will be summed and divided by 6 to calculate the average PD for each patient.
clinical attachment level | During the first 1 day visit
  With the help of a periodontal probe, the distance between the enamel-cement border and the sulcus/pocket base will be measured at six points of the tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatinal/lingual, mid buccal/palatinal and distobuccal/palatinal. The values will be summed and divided by 6 to calculate the average amount of clinical attachment level for each patient.
plaque index | During the first 1 day visit
  For Silness&Löe plaque index measurement, values will be obtained from four surfaces of each tooth: mesial, distal, vestibular and palatinal. The values will be summed and divided by four to determine the PI score for each tooth. Scoring will be done as follows; 0: No bacterial plaque on the gingival area of the tooth surface. 1: No bacterial plaque is visible on the surface of the tooth by eye, but after probing, bacterial plaque is observed at the tip of the probe. 2: The gingival area is covered with a thin to moderate amount of bacterial plaque, which is visible by eye. 3: There is a large amount of soft debris, the thickness of which completely fills the gingival groove and the interdental space is filled with soft debris.
gingival index | During the first 1 day visit
  According to Löe&Silness gingival index; vestibule, lingual, mesial and distal surfaces of all teeth will be examined. The values will be summed and divided by four to determine the GI score for each tooth. 0: Healthy gingiva. 1: Mild inflammation, mild discoloration and edema but no bleeding after probing. 2: Moderate inflammation, edema, redness and brightness, bleeding on probing. 3: Severe inflammation and redness, edema, ulceration and tendency to spontaneous bleeding.
bleeding on probing | During the first 1 day visit
  The following index criteria will be used to determine the degree of inflammation in the soft tissue surrounding the vestibular, lingual, mesial and distal surfaces of all teeth. The number of positive (+) scoring areas on the examined surfaces will be calculated as a percentage of the total number of examined areas. (-): No bleeding when the periodontal probe is passed along the gingival sulcus. (+): Bleeding is present at the gingival margin.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir Katip Celebi University Faculty of Dentistry, Izmir, Cigli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No